CLINICAL TRIAL: NCT06125210
Title: Application of Early Bundle Management of Mechanical Ventilation to Prevent Ventilator Dependence in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: fdpicu-25
Record Dates: First submitted 2023-11-06; First posted 2023-11-09 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Prolonged Mechanical Ventilation
MeSH Terms: interventions — Food Assistance; Tracheotomy

STUDY DESIGN:
Intervention Model Description: Intervention group: The bundle treatment plan was:1) After receiving mechanical ventilation for <7 days, three of the following four items of intensive bedside rehabilitation were initiated: ① electrical diaphragm stimulation, ② electrical muscle stimulation, ③ passive limb movement, ④ respiratory rehabilitation.
  2) Receive mechanical ventilation <14 days, start the target-oriented nutrition program, including: (1) nutrition department consultation, (2) MDT to develop individualized nutritional pathways, nutrient formulations and use methods, and achieve the target nutritional level within 2 weeks.
  3) Receiving mechanical ventilation <21 days, tracheotomy transition to home mechanical ventilation (HMV), special diseases (central nervous system diseases) receiving mechanical ventilation 14-21 days recommended tracheotomy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Behavioral: early bedside rehabilitation; Dietary Supplement: nutrition program; Procedure: tracheotomy
- control group (No Intervention)

INTERVENTIONS:
Behavioral: early bedside rehabilitation — ① electrical diaphragm stimulation, ② electrical muscle stimulation, ③ passive limb movement, ④ respiratory rehabilitation.
  Arms: intervention group
Dietary Supplement: nutrition program — (1) nutrition department consultation, (2) MDT to develop individualized nutritional pathways, nutrient formulations and use methods, and achieve the target nutritional level within 2 weeks
  Arms: intervention group
Procedure: tracheotomy — early tracheotomy for special diseases (e.g central nervous system diseases) receiving mechanical ventilation 14-21 days recommended tracheotomy
  Arms: intervention group

SUMMARY:
This study is based on the risk factors of previous studies to formulate a bundle treatment plan to prevent ventilator dependence in children, in order to reduce the proportion of ventilator dependence in children and provide a theoretical basis for reasonable intervention of children with mechanical ventilation.

Participants will receive intensive rehabilitation, nutrition, and tracheotomy at different time periods.

Researchers will compare the control group to see whether it can reduce the incidence of ventilator dependence

ELIGIBILITY:
Inclusion Criteria:

（1）All stable children receiving mechanical ventilation

（1）Stable condition: respiratory rate does not exceed 20% of the basic respiratory rate, PEEP< 8. 60%, VIS score< 20, there is no hypotension (70mmHg+ age ×2, 70mmHg under one year old), no higher than the P95 of the same sex and age

Exclusion Criteria:

1. Status epilepticus
2. Active intracranial hemorrhage
3. Intracranial hypertension
4. Unstable fracture of the spine
5. Spinal cord injury
6. There are injuries that affect the implementation of rehabilitation
7. Acute surgery was performed on the same day.
8. Body temperature over 40℃
9. Brain function failure

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
limb skeletal muscle function indexes | 21 days after enrollment
  Skeletal muscle thickness and cross-sectional area were measured

CONTACTS AND LOCATIONS:
Locations (1):
- Children's hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No